CLINICAL TRIAL: NCT02742558
Title: A Randomized Observer Blinded Controlled Non Inferiority Trial to Evaluate the Safety and Immunogenicity of Locally Manufactured Inactivated Bivalent Whole Cell-oral Cholera Vaccine (WC-OCV) 'Cholvax' in Bangladeshi Healthy Adults and Children
Brief Title: Safety and Immunogenicity of Locally Manufactured Oral Cholera Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: International Vaccine Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PR-15076
Record Dates: First submitted 2016-04-07; First posted 2016-04-19 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2016-10

CONDITIONS: Cholera
Keywords: cholera vaccine; randomized trial; immunogenicity
MeSH Terms: conditions — Cholera | interventions — shanchol

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cholvax (Experimental): Incepta vaccine Limited, a leading pharmaceutical company in Bangladesh is now producing the OCV, Cholvax with technological support from International Vaccine Institute (IVI), which meets international Good Manufacturing Practice (GMP) standards and WHO production guidelines. Cholvax has the same formulation as ShancholTM in terms of strains and formulation.
  Interventions: Biological: Cholvax
- shanchol (Active Comparator): The vaccine is manufactured by Shantha Biotechnics, in Hyderabad, India and is prequalified by the WHO. Shanchol™ is available in a single dose vial.This vaccine is used as two dose regimen.
  Interventions: Biological: Shanchol

INTERVENTIONS:
Biological: Cholvax — Incepta vaccine Limited, a leading pharmaceutical company in Bangladesh is now producing the OCV, Cholvax with technological support from International Vaccine Institute (IVI), which meets international Good Manufacturing Practice (GMP) standards and WHO production guidelines. Cholvax has the same formulation as ShancholTM in terms of strains and formulation.
  Arms: cholvax
Biological: Shanchol — The vaccine is manufactured by Shantha Biotechnics, in Hyderabad, India and is prequalified by the WHO. Shanchol™ is available in a single dose vial.This vaccine is used as two dose regimen.
  Arms: shanchol

SUMMARY:
To evaluate and compare the safety and immunogenicity of the Cholvax with ShancholTM, Investigators will conduct a clinical trial study Bangladeshi healthy adults and children. Cholvax is locally produced orally administered whole cell inactivated bivalent cholera vaccine. Incepta vaccine Limited, a leading pharmaceutical company in Bangladesh is now producing the oral cholera vaccine, Cholvax with technological support from International Vaccine Institute (IVI). Cholvax meets international Good Manufacturing Practice (GMP) standards and WHO production guidelines. Cholvax has the same formulation as ShancholTM in terms of strains and formulation. By this transfer of technology, it expected that the vaccine will become available for use in public health programs in Bangladesh and in the future in other cholera-affected countries in Asia and Africa to control endemic cholera, as well as to help control large-scale epidemics and outbreaks.

Investigators will also evaluate and compare the safety and immunogenicity of 3 Cholvax lots (lot-to-lot consistency).

DETAILED DESCRIPTION:
Background : Cholera continues to be a major cause of morbidity and mortality in low-income countries including Bangladesh. It is estimated that there are at least 300,000 severe cases and over 4,500 deaths in Bangladesh each year1. The overall morbidity for cholera remains high. A global stockpile of OCV has been created by WHO in 2013 for epidemic and outbreak settings2. However, the global demand for the vaccine far exceeds the present supply for both epidemic and also endemic settings3. It can be envisioned that local production of an affordable OCV for high risk population in endemic settings will improve the present scenario in Bangladesh and other countries.

Knowledge gap: The WHO recommends OCV for use in both endemic and epidemic cholera settings4. At present there are two vaccines that are WHO prequalified. These include Dukoral which is registered in Bangladesh and in over 50 countries. However, the disadvantage of use of Dukoral is that its current price it is expensive for Bangladesh and other developing countries. In addition, the need for buffer to formulate the vaccine makes it less fieldable for mass vaccination programs. Another whole cell killed OCV, ShancholTM, which is WHO prequalified, is based on similar bacterial components as Dukoral and licensed in India but not in Bangladesh. Although this vaccine is relatively affordable it may not be sufficiently cost effective for the Government of Bangladesh to implement it in our poor endemic settings. At present, the vaccine is in short supply and will not be able to meet the global demands. In order to increase supply of OCV and make the vaccine more affordable, a locally manufactured killed bivalent whole cell-oral cholera vaccine Cholvax is now available. The present study will evaluate the safety and immunogenicity of Cholvax as a test vaccine using Shanchol TM as the comparator vaccine in a non inferiority trial design.

Relevance: The study of this locally manufactured OCV, Cholvax among children and adults will be able to give us information regarding the safety and immunogenicity of the vaccine. Based on this information, it can be anticipated that regulatory requirements as well as licensure of the vaccine will be initiated in Bangladesh. This will pave the way forward for the future approval by WHO and for its global use. The introduction of Cholvax in endemic settings, seasonal outbreak as well as in the EPI program of the country in the future can be expected based on the study results; initiatives and plans can be made to introduce this locally produced vaccine in Bangladesh at an affordable cost and in the future globally.

Hypothesis (if any): Locally produced orally administered whole cell inactivated bivalent cholera vaccine, Cholvax is non inferior or at least as safe and immunogenic in adults and children in Bangladesh as compared to Shanchol TM.

Objectives: The objectives of this study are- i. To evaluate and compare the safety and immunogenicity of the Cholvax with ShancholTM ii. To evaluate the safety and immunogenicity of Cholvax in healthy adults and children in Dhaka.

iii. To evaluate and compare the safety and immunogenicity of 3 Cholvax lots (lot-to-lot consistency) Methods: This will be a randomized, observer blinded and comparative study on a total of 2052 healthy participants, 1026 Cholvax (Test Group) and 1026 ShancholTM (Comparator Group) recipients. There will be three age cohort arms in each test and comparator group which will consist of 219 participants for age 1-5Yrs, 373 participants for age 6-17Yrs and 434 for Age 18-45Yrs, with a total of 2052 participants. Participants will receive either Cholvax or ShancholTM two doses 14 days apart.

Each age cohort of the study (Cohort I onwards) will be completed and based on the development, and progress, the next age cohort will be initiated. If the vaccine is found to be safe in the adults it will be tested in the children, 6-17 years of age and followed by the younger age group 1-5 years of age. The results will be presented to the Data Safety Monitoring Board after completing the 28-day safety surveillance part of each age cohort of the study and before proceeding to the next study age cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 1-45 Years.
2. Informed consent from study participants and guardian in case of children (1-17 years) and assent from children aged 11-17 years.
3. Participation in the study at least for next 6 months
4. Considered healthy as per medical judgment of the investigator

Exclusion Criteria:

1. Suffering from diarrhea or abdominal pain or vomiting in the past 24 hours or diarrhea lasting for more than 2 weeks in the past 6 months
2. History of taking oral cholera vaccine and history of confirmed cholera.
3. History of taking any other live or killed enteric vaccine in the last 8 weeks.
4. History of anaphylaxis or serious vaccine reaction.
5. Currently use of any immunosuppressive or immune-modifying drugs. 6.100.4 0 F (38℃) or higher body temperature measured prior to investigational product dosing.

7.Receipt of blood or blood products or parenteral immunoglobulin preparation in the past 3 months.

8.Currently on antimicrobial therapy. 9.Severe malnutrition or chornic disease based on the jugement of the investigator.

10.Stool sample at screening positive for V. cholerae. 11.Pregnant women or plans to become pregnant during the study period .

Ages: 1 Year to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2052 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with vaccine related reactogenicity as assessed by study personnel | Within 30 minutes after administration of vaccine
  Number of reactogenecity events will be compared between test group and comparator group.
Number of participants with solicited adverse events as assessed by study personnel | Within 7 days after administration of vaccine
  Number of solicited adverse events observed after each dose of vaccination assessed by study personnel through home visit and will be compared between test group and comparator group
Number of participants with unsolicited adverse event including serious adverse event as assessed by study physician | Within 6 months after administration of vaccine
  Number of unsolicited adverse events including serious adverse event observed after each dose of vaccination assessed by study personnel through home visit and will be compared between test group and comparator group
Number of participants showing seroconversion against sero group V. cholerae O1 | 7 days after administration of vaccine
  Proportion of participants showing sero-conversion against V. cholerae O1, upon vaccination Cholvax being tested in comparison with ShancholTM.

SECONDARY OUTCOMES:
Number of participants showing seroconversion against sero group V. cholerae O139 | 7 days after administration of vaccine
  Proportion of participants showing sero-conversion against serogroup V. cholerae O139 upon vaccination with Cholvax in comparison with ShancholTM will be measured and compared between test and comparator group Geometric Mean Titer (GMT) and Geometric Mean Ratio (GMR) as measured by anti-V. cholerae O1 antibody titer at day 7 and day 21 after the first dose of investigational product dose as compared to baseline (day0).
  Geometric Mean Titer (GMT) and Geometric Mean Ratio (GMR) as measured by anti-V. cholerae O139 antibody titer at day 7 and day 21 after the first dose of investigational product dose as compared to baseline (day 0).

CONTACTS AND LOCATIONS:
Overall Officials: Firdausi Qadri, Dr., Study Director — International Centre for Diiarrhoeal Disease Research, Bangladesh
Locations (1):
- International Centre for Diarrhoeal Disease Research, Bangladesh, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with International Vaccine Institute

REFERENCES:
- [Result] Ali M, Lopez AL, You YA, Kim YE, Sah B, Maskery B, Clemens J. The global burden of cholera. Bull World Health Organ. 2012 Mar 1;90(3):209-218A. doi: 10.2471/BLT.11.093427. Epub 2012 Jan 24. PMID 22461716
- [Result] Maskery B, DeRoeck D, Levin A, Kim YE, Wierzba TF, Clemens JD. Strategy, demand, management, and costs of an international cholera vaccine stockpile. J Infect Dis. 2013 Nov 1;208 Suppl 1:S15-22. doi: 10.1093/infdis/jit233. PMID 24101640
- [Result] Saha A, Chowdhury MI, Khanam F, Bhuiyan MS, Chowdhury F, Khan AI, Khan IA, Clemens J, Ali M, Cravioto A, Qadri F. Safety and immunogenicity study of a killed bivalent (O1 and O139) whole-cell oral cholera vaccine Shanchol, in Bangladeshi adults and children as young as 1 year of age. Vaccine. 2011 Oct 26;29(46):8285-92. doi: 10.1016/j.vaccine.2011.08.108. Epub 2011 Sep 9. PMID 21907255